CLINICAL TRIAL: NCT00827008
Title: An Open-Label, Long-Term Treatment Study to Assess the Long-Term Safety and Tolerability and Efficacy of Neramexane With Subjective Tinnitus
Brief Title: Open-Label, Long-Term Treatment Study, to Assess the Long-Term Safety and Tolerability and Efficacy of Neramexane in Patients With Subjective Tinnitus
Acronym: OLLTT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRZ 92579/TI/3004; 2008-001432-13 (EudraCT Number)
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Subjective Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1, verum (Experimental)
  Interventions: Drug: Neramexane mesylate

INTERVENTIONS:
Drug: Neramexane mesylate — Up-titration treatment period of 5 weeks up to 75mg Neramexane mesylate oral per day followed by 49 weeks treatment maintenance

SUMMARY:
The purpose of this study is to investigate the long-term safety and tolerability and efficacy of neramexane mesylate in the long-term treatment of subjective tinnitus after a completed double-blind randomized placebo controlled study

ELIGIBILITY:
Main Inclusion Criteria:

* Male or female patients who have successfully completed one of the double-blind Phase 3 tinnitus studies of Merz with Neramexane mesylate
* patients aged equal or older 18 but not older than 75 years with clinical diagnosis of first onset, persistent (i.e. tinnitus should never be absent for more than 24 hours in a row), subjective, uni-or bilateral subacute tinnitus at the timepoint of the lead-in study

Main Exclusion Criteria:

* clinical diagnosis of intermittent or pulsatile tinnitus
* Patients who have tinnitus as a concomitant symptom of an otological/neurological disease (such as otitis media, Meniére´s disease, otosclerosis etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 821 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Descriptive analyses of TBF-12 (Tinnitus-Beeinträchtigungs-Fragebogen 12 "Tinnitus Handicap Inventory 12")total score and its subscores, of the Tinnitus Rating Scale and its single items as well as of SF-36 and safety/tolerability parameters | 54 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — Merz Pharmaceuticals
Locations (134):
- United States (30):
  - Paradigm Clinical Research, Tucson, Arizona
  - Providence Clinical Research, Burbank, California
  - Central California Clinical Research, Fresno, California
  - UC Davis Health System Department of Otolaryngology, Sacramento, California
  - Colorado Otolaryngology Associates, Colorado Springs, Colorado
  - New West Physicians, Golden, Colorado
  - Visions Clinical Research, Boynton Beach, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Deerpath Physicians Group, Gurnee, Illinois
  - Knight Center for Integrated Health,, Peoria, Illinois
  - University of Kansas Department of Otolaryngology Head & Neck Surgery, Kansas City, Kansas
  - Heartland Research Associates, LLC., Wichita, Kansas
  - Commonwealth Ear, Nose & Throat, Louisville, Kentucky
  - Glacier Ear, Nose, and Throat, Head and Neck Surgery, P.C., Kalispell, Montana
  - Immedicenter, Bloomfield, New Jersey
  - David L. Bortniker, M.D, FACS, Somerville, New Jersey
  - Erie County Medical Center, Department of Rehabilitation Medicine, Buffalo, New York
  - Montefiore Medical Center Attn: Anxiety and Depression Center, The Bronx, New York
  - Cary Medical Research, Cary, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Wilmington Medical Research, Wilmington, North Carolina
  - Piedmont Medical Research, Winston-Salem, North Carolina
  - Medical University of South Carolina - Department of Otolaryngology, Department of Otolaryngology - Head & Neck Surgery, Charleston, South Carolina
  - Future Search Trials of Neurology, Austin, Texas
  - FutureSearch Trials of Dallas, Dallas, Texas
  - R/D Clinical Research, Inc., Lake Jackson, Texas
  - South Texas Research Alliance LLC, Laredo, Texas
  - Research Across America, Plano, Texas
  - Advanced Clinical Research, West Jordon, Utah
  - Health Research of Hampton Roads, Inc., Newport News, Virginia
- Austria (3):
  - Krankenhaus der Elisabethinen, Graz
  - Bezirkskrankenhaus Kufstein Dr. Christof Pauli (PI: Prim. Dr. Peter Ostertag, Kufstein
  - Clin Pharm International GmbH, Zentrum Wien, Vienna
- Belgium (4):
  - University Hospital Brussels, Brussels
  - Clinique Universitaire Saint-luc, Brussels
  - AZ Sint Lucas, ENT department, Ghent
  - University Hospital Leuven, ENT Department, Leuven
- Brazil (4):
  - Consultório Dr. Marcelo Rates, Belo Horizonte/Mimaf Gerais
  - Osmar Clayton Person, Santo André/SP
  - Instituto Ganz Sanchez, São Paulo/SP
  - Clínica OTOSUL, Valenca/RJ
- Czechia (8):
  - Medico, Chodov, Prague
  - prof. MUDr. Ivo Šlapák, Brno
  - Teaching University Hospital, ORL klinika, Brno
  - ORL oddělení, Karlovarská krajská nemocncie a.s., Karlovy Vary
  - Oblastní nemocnice Kladno a.s., Nemocnice Středočeského kraje, Kladno
  - Pro-audio,s.r.o.-private ENT clinic, Mladá Boleslav
  - ORL oddělení, Všeobecná Fakultní Nemocnice v Praze, Prague
  - ORL oddělení , Karlovarská krajská nemocnice a. s., Sokolov
- France (9):
  - Dr. Ebbo, Issy-les-Moulineaux
  - Dr. Sarfati, La Seyne-sur-Mer
  - Centre Hospitalier de Bretagne Sud Service ORL-B9, Lorient
  - Dr. Bonfils, Paris
  - Dr. Ohresser, Paris
  - Hopital Nord, Saint-Etienne
  - Dr. Fraysse, Toulouse
  - Service ORL CHU Bretonneau, Tours
  - Hopital Paul BROUSSE Polyclinique, Villejuif
- Germany (21):
  - Dr. Kühne, Elisabeth, Halle, Saale
  - Dr. med. Norbert Pasch, Aachen
  - Charité, Universitätsmedizin Berlin-Tinnituszentrum, Berlin
  - Klin. Forschung Berlin Buch GmbH, Berlin
  - Dr. med. Frank Reintjes, Braunschweig
  - DM Helena Sigal, Chemnitz
  - Dr. Klaus Peter Jayme, Darmstadt
  - Dr. Christian Dörr, Dresden
  - HNO-Praxis im Gesundheitszentrum, Duisburg
  - Dr. Gieselmann, Werner, Heiligenhaus
  - Dr. Wolfgang Lotte, Iserlohn
  - Dr. Dr. med. Hans-Detlev Stahl, Leipzig
  - HNO Praxis, Lichtenfels
  - Dr. Dannesberger, Lorsch
  - ClinPharm International, Magdeburg
  - HNO Gemeinschaftpraxis, Meppen
  - Martin Canis, MD, Munich
  - Dr. med. Ulrike Walter, Nuremberg
  - Dr. Susanne Wiedemann, Nuremberg
  - Dr. Norbert Staab, Schlüchtern
  - Dr. Hannelore Neumaier, Wiesbaden
- Mexico (12):
  - Unidad Médica de Especialidades del Noroeste (UMEN), Centro Culiacán Sinaloa
  - Hospital General de Chihuahua. "Dr. Salvador Anchondo", Chihuahua C.P. 31000
  - Hospital Christus Muguerza del Parque, Chihuahua CP 3100
  - Internal Medicine Clin Trials (IMED), Col Obispado, Monterrey , N.L. C.P. 64060
  - Hospital Civil de Guadalajara, Col. El Retiro CP 44280 Cuadalajara Jalis
  - Grupo Médico Terranova, CP 44630 Guadalajara Jalisco
  - Clinical Research Instutute S.C., Edo. de México CP 54055
  - Instituto Biomédico de Investigación A.C., Fracc. Bosques Del Prado Norte Aguascalientes
  - Unidad de Investigación Clínica Cardiometábolica de Occidente S.C. (UNICAMO), Jalisco
  - Monterrey International Research Center (MIRC), Nuevo León CP 64000
  - Hospital Universitario Dr. José Eleuterio González. Edificio Elizondo Barragán, Servicio de Otorrinolaringología, Nuevo León CP 64400
  - Hospital Central "Dr. Ignacio Morones Prieto" Servicio de Otorrinolaringología, San Luis Potosí, SLP, México, 78240
- Netherlands (7):
  - Andromed Zoetermeer, Zoetermeer, EK
  - Andromed Oost, Velp, ES
  - Rijnland Ziekenhuis, ENT department, Leiderdorp, GA
  - Andromed Rotterdam, Rotterdam, HC
  - Adromed Nijmegen, Nijmegen, HL
  - Andromed Leiden, Leiderdorp, RA
  - Andromed Breda, Breda, VL
- Poland (13):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Niepubliczny Zaklad Opieki Zdrowotnej Prywatne Centrum Medyczne PROMEDIS, Gdansk
  - Szpital Miejski im. J.Brudzinskiego, Gdynia
  - Samodzielny Publiczny Szpital Kliniczny im. Andrzeja Mieleckiego Slaskiego Uniwersytetu Medycznego w Katowicach, Katowice
  - NZOZ Specjalistyczne Centrum Medyczne Nowomed, Krakow
  - Niepubliczny Zaklad Opieki Zdrowotnej PROMED, Krakow
  - Specjalistyczny Gabinet Otolaryngologiczny, Krakow
  - Szpital Specjalistyczny im. Stefana Zeromskiego, SP ZOZ w Krakowie, Oddzial Otolaryngologii, Krakow
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej, Uniwersytecki Szpital Kliniczny nr 1 im. Norberta Barlickiego Uniwersytetu Medycznego w Lodzi, Lodz
  - Wojewodzki Szpital Specjalistyczny im. Stefana Kardynała Wyszynskiego Samodzielny Publiczny Zaklad Opieki Zdrowotnej, Lublin
  - Wojewodzki Szpital Specjalistyczny w Olsztynie, Olsztyn
  - Instytut Fizjologii i Patologii Sluchu, Warsaw
  - Samodzielny Publiczny Szpital Kliniczny nr 1 we Wroclawiu, Wroclaw
- Hospital Militar Regional nº 1 Serviço de Otorrinolaringologia, Porto, Portugal
- South Africa (6):
  - Louis Leipoldt Mediclinic, Bellville
  - Lakeview Hospital, Benoni
  - 1007 Louis Pasteur Building, Pretoria
  - GCT Eastmed Clinical Trial centre, Pretoria
  - Constantiaberg Medi Clinic,, Western Cape
  - Prince Alfred House, Wynberg
- Spain (7):
  - Hospital Sagunto, Sagunto, Valencia
  - Fundación Hospital de Alcorcón, Otorhinolaryngology, Alcorcon - Madrid
  - Hospital Clínico Barcelona, Dept. Of ORL, Barcelona
  - Hospital Puerta del Hierro, Madrid- Servicio de ORL, Madrid
  - Hospital Universitario Príncipe de Asturias, Madrid
  - Clínica Universitaria de Navarra, Dept. ORL, Pamplona, Navarra
  - Hospital Universitario de Salamanca- Hospital Virgen de la Vega, Salamanca
- United Kingdom (9):
  - Oldfield Surgery, Bath
  - Addenbrooke's Hospital, Cambridge
  - Avondale Surgery, Research Office, Chesterfield
  - The university Hospitals of Leicester, Leicester Royal Infirmary, Leicester
  - Burbage Surgery, Leicestershire
  - The Freeman Hospital, Newcastle upon Tyne
  - Wansford and Kings Cliffe Practice, Petereborough
  - Frome Medical Practice, Somerset
  - Sherbourne Medical Centre, Warwickshire